CLINICAL TRIAL: NCT05952141
Title: Thibang Diphatlha: Testing Adaptive Strategies to Close the Gap From Cervical Cancer Diagnosis to Treatment in Botswana
Brief Title: Strategies to Close the Gap From Cervical Cancer Diagnosis to Treatment in Botswana
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Botswana (Other)
Responsible Party: Principal Investigator, Katharine Rendle, Principal Investigator, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: UPCC 23822; U01CA275032-01 (NIH)
Record Dates: First submitted 2023-07-11; First posted 2023-07-19 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer
Keywords: Screening; Botswana; Treatment; Patient
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Pragmatic Sequential Multiple Assignment Randomized Trial (SMART).
  This study uses a sequential randomization design in which all eligible participants will be randomized into one of two interventions at Stage 1 and then participants that do not respond to Stage 1 interventions will be randomized to receive Stage 2 interventions
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1 Clinic Outreach + Stage 2 Low Touch (Experimental): All participants receive direct clinic outreach to communicate readiness of results (stage 1). Participants who do not attend the clinic by 30 days (non-responders) will receive asynchronous text message reminders using framed messaging (stage 2).
  Interventions: Behavioral: Clinic Outreach; Behavioral: Low-Touch Strategy
- Stage 1 Clinic Outreach + Stage 2 High Touch (Experimental): All participants receive direct clinic outreach to communicate readiness of results (stage 1). Participants who do not attend the clinic by 30 days (non-responders) will receive asynchronous text message reminders using framed messaging in combination with synchronous patient navigation (stage 2).
  Interventions: Behavioral: Clinic Outreach; Behavioral: High-Touch Strategy
- Stage 1 Enhanced Outreach + Stage 2 Low-Touch (Experimental): All participants receive direct clinic outreach plus enhanced outreach to communicate readiness of results (stage 1). Participants who do not attend the clinic by 30 days (non-responders) will receive asynchronous text message reminders using framed messaging (stage 2).
  Interventions: Behavioral: Enhanced Outreach; Behavioral: Low-Touch Strategy
- Stage 1 Enhanced Outreach + Stage 2 High-Touch (Experimental): All participants receive direct clinic outreach plus enhanced outreach to communicate readiness of results (stage 1). Participants who do not attend the clinic by 30 days (non-responders) will receive asynchronous text message reminders using framed messaging in combination with synchronous patient navigation.
  Interventions: Behavioral: Enhanced Outreach; Behavioral: High-Touch Strategy

INTERVENTIONS:
Behavioral: Clinic Outreach — A member of the pathology team will contact the referring clinic to communicate the readiness of results.
  Arms: Stage 1 Clinic Outreach + Stage 2 High Touch; Stage 1 Clinic Outreach + Stage 2 Low Touch
Behavioral: Enhanced Outreach — A member of the pathology team will contact both the referring clinic and the patient directly to communicate the readiness of results.
  Arms: Stage 1 Enhanced Outreach + Stage 2 High-Touch; Stage 1 Enhanced Outreach + Stage 2 Low-Touch
Behavioral: Low-Touch Strategy — Patient will be sent asynchronous text messaging reminders related to the importance of timely care using framed messaging.
  Arms: Stage 1 Clinic Outreach + Stage 2 Low Touch; Stage 1 Enhanced Outreach + Stage 2 Low-Touch
Behavioral: High-Touch Strategy — Patient will be sent asynchronous text messaging reminders related to the importance of timely care using framed messaging in combination with synchronous telephone-based patient navigation.
  Arms: Stage 1 Clinic Outreach + Stage 2 High Touch; Stage 1 Enhanced Outreach + Stage 2 High-Touch

SUMMARY:
Investigators will test the effectiveness of adaptive strategies on timely adoption of cervical cancer treatment in Botswana using a pragmatic trial design.

DETAILED DESCRIPTION:
Investigators will test the effectiveness of adaptive strategies on timely adoption of cervical cancer treatment in Botswana using a hybrid (type III) and pragmatic Sequential Multiple Assignment Randomized Trial (SMART) design. The adaptive strategies are designed to target patient- and system-level determinants identified in preliminary data, including delayed communication of results, individual and structural barriers to accessing treatment, and suboptimal care coordination between referring and cancer treatment clinics. The strategies draw upon key principles in behavioral economics and are supported by systematic evidence of the effectiveness of nudge strategies in preventive, HIV, and cancer care. The overarching rationale for the study is that enhancing coordination, communication, and navigation through centralized outreach and nudge strategies will increase timely treatment adoption and be scalable and sustainable in the long-term.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible if they:

1. are biological females
2. are aged 18 or older
3. have pathology-confirmed invasive cervical cancer diagnosis
4. have pathology results evaluated at National Health Laboratory in Botswana
5. are citizens of Botswana
6. have no prior history of invasive cervical cancer

Exclusion Criteria:

Patients will be excluded if they:

1. are biological males or otherwise born without a cervix
2. are below the age of 18 due to the rarity of cervical cancer in this population
3. do not meet study inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Adoption | Within 90 days of randomization
  Defined as the initiation of cervical cancer treatment within 90 days of randomization.

SECONDARY OUTCOMES:
Fidelity | 12 months after randomization
  Defined as completion of evidence-based cancer treatment according to international guidelines and measured using medical record data.
Reach: First Appointment | 12 months after randomization
  Defined by the proportion of patients who complete an initial treatment visit divided by those randomized
Reach: First Stage | 12 months after randomization
  Defined by the proportion of patients who complete an enhanced outreach phone call divided by those contacted.
Reach: Second Stage | 12 months after randomization
  Defined by the proportion of patients who complete a patient navigation phone call (high touch strategy) divided by those contacted.
Reach: Results | 12 months after randomization
  Defined by the proportion of patients with confirmation of results received divided by those randomized.

OTHER OUTCOMES:
Clinical Outcomes: Treatment | 12 months after randomization
  Defined by the stage at diagnosis, type of cancer treatment the patient received (e.g., chemoradiation, surgery) measured using medical record data.
Clinical Outcomes: Survival | 12 months after randomization
  Defined as overall survival at one year after randomization measured using medical record data.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Rendle, PhD,MSW,MPH, Principal Investigator — University of Pennsylvania; Surbhi Grover, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (3):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Botswana (2):
  - Nyangabgwe Referral Hospital, Francistown, North-East District
  - Princess Marina Hospital, Gaborone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rendle KA, Ramogola-Masire D, Grover S; Thibang Diphatlha Collective. Thibang Diphatlha: a sequential multiple assignment randomized trial designed to increase timely adoption of cervical cancer treatment in Botswana. Implement Sci Commun. 2024 Nov 12;5(1):128. doi: 10.1186/s43058-024-00659-9. PMID 39533437